CLINICAL TRIAL: NCT03294070
Title: A 24-week Open-label Clinical Trial to Assess Tolerability and Antihypertensive Effect and in Hemodynamic Parameters and Arterial Stiffness of Fimasartan 60 mg Plus Amlodipine Besylate 5 mg Given Once a Day in Patients With Hypertension in Stadiums 2/3
Brief Title: Fimasartan Plus Amlodipine on Hemodynamic Parameters and Arterial Stiffness in Patients With Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Ernesto German Cardona Muñoz, Ernesto German Cardona Muñoz, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTEC-1
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Arterial Hypertension
Keywords: hemodynamic parameters; arterial stiffness
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fimasartan 60 mg + amlodipine besylate 5 mg (Experimental): Fimasartan 60 mg + amlodipine besylate 5 mg. In subjects with a DBP equal to or greater than 90 mmHg and / or SBP equal to or greater than 140 mmHg at week 8, the investigator will have the option, according to his clinical criteria, to add 12.5 mg of HCTZ QD (in these cases, the subject will receive one 60 mg Fimasartan tablet plus 12.5 mg HCTZ plus one 5 mg amlodipine besylate tablet.
  Interventions: Combination Product: Fimasartan plus amlodipine besylate

INTERVENTIONS:
Combination Product: Fimasartan plus amlodipine besylate — Fimasartan 60 mg plus amlodipine besylate 5 mg or Fimasartan plus 12.5 mg HCTZ plus one 5 mg amlodipine besylate

SUMMARY:
24-week open clinical trial to assess tolerability and effect on pressure, hemodynamic parameters and arterial rigidity of the combined treatment based on Fimasartan 60 mg and amlodipine besylate 5 mg given once daily in patients with arterial hypertension in stages 2-3

DETAILED DESCRIPTION:
A prospective, open clinical trial of a cohort of adult patients of both sexes with recent 2-3 years high blood pressure.

Intervention: Fimasartan 60 mg + amlodipine besylate 5 mg once daily

Purpose and justification of the study:

Systemic arterial hypertension (SAH) is a pathology that diminishes the hope and quality of life and is directly associated with the production or aggravation of other pathologies such as atherosclerosis, heart failure, ischemic heart disease and / or chronic kidney disease.

Several studies have shown that central pulse pressure (cPP) and central aortic pressure (CAP) are better predictors of cardiovascular disease, target organ damage and mortality, than the brachial or peripheral pulse pressure (pPP). More attention should be paid to central hemodynamics, since its values are those that directly impact the organs that are commonly damaged as a result of hypertension, brain, kidney and heart. (2) Current therapeutic strategies for SH, although partially effective, have not adequate control of tension figures in hypertensive patients, either due to lack of power, by their adverse effects or by requiring multiple shots that seriously compromise attachment to the treatment. Fimasartan is a medicine that belongs to the therapeutic class of the selective blockers of angiotensin II (AT 1) receptors, family of drugs with less adverse effects than other renin-angiotensin-aldosterone axis inhibitors, with potency adequate antihypertensive and additional beneficial effects on renal function, hypertrophy ventricular, atheromatosis and insulin sensitivity. Based on the physico-chemical characteristics of the Fimasartan and the results obtained in phase I-II and III studies in different populations, including the Mexican,favoring the adherence and control of blood pressure, it can be an effective and safe therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

1. Subject capable of understanding and signing voluntarily informed consent.
2. Men and women aged 18-65 years.
3. To have essential hypertension grade 2 or 3 according to the figures of diastolic blood pressure and / or systolic in office according to NOM-030 SSA.
4. Reliable and willing to attend all study visits for the duration of the study and the follow-up according to the researcher's criteria.
5. Patients on antihypertensive treatment and who in the judgment of the investigator and taking care of the health and safety of the patient can undergo 2 weeks of previous washing to the visit of day 0.

   -

Exclusion Criteria:

1. Secondary arterial hypertension.
2. Patients currently under treatment that at the discretion of the investigator can not be submitted to wash period.
3. Severe renal insufficiency (glomerular filtration rate <30 mL / min / 1.73 m2)
4. Moderate to severe hepatic impairment (Child-Pugh B or C classification).
5. Hypersensitivity to any of the components of the research products
6. Hepatobiliary obstruction
7. Myocardial infarction or severe coronary artery disease (including angina pectoris unstable) or clinically significant congestive heart failure within 6 months prior to visit to week-1 (selection).
8. Left ventricular ejection fraction ≤40%
9. Resting heart rate ≥90 lpm
10. Thyroid disorder (treated subjects may be involved who are euthyroid)
11. Clinically significant mitral or aortic valve disease (Grade ≥ 2) Hypertrophic obstructive cardiomyopathy

13. Clinically significant rhythm disorders 14. Clinically significant abnormal laboratory parameters in the investigator's judgment.

15. Concurrent treatment that may affect blood pressure and which can not be withdrawn in the opinion of the investigator. 16. A history of galactose intolerance or glucose-galactose malabsorption. 17. Pregnancy, breastfeeding. 18. Women capable of procreation DO NOT adopt an effective contraceptive method according to criterion of the investigator.

19. Patients participating in or participating in other research protocols within 3 months prior to week 1 visit (selection). 20. Another reason not previously specified but in the opinion of the investigator may contraindicate their participation in the study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Reduction of pulse wave velocity | 24 week
  The administration of combined dose-based treatment of 60 mg of fimasartan plus 5 mg of amlodipine besylate QD administered according to the treatment schedule for 24 weeks reduces VOPcf in Mexican Patients with Essential Arterial Hypertension grades 2 and 3

SECONDARY OUTCOMES:
Central Aortic Pressure | 24 week
  The administration of combined dose-based treatment of 60 mg of fimasartan plus 5 mg of amlodipine besylate QD administered according to the treatment schedule for 24 weeks reduces Central Aortic Pressure in Mexican Patients with Essential Arterial Hypertension grades 2 and 3
Central Pulse Pressure | 24 week
  The administration of combined dose-based treatment of 60 mg of fimasartan plus 5 mg of amlodipine besylate QD administered according to the treatment schedule for 24 weeks reduces Central Pulse Pressure in Mexican Patients with Essential Arterial Hypertension grades 2 and 3
Rising Index | 24 week
  The administration of combined dose-based treatment of 60 mg of fimasartan plus 5 mg of amlodipine besylate QD administered according to the treatment schedule for 24 weeks reduces Rising Index in Mexican Patients with Essential Arterial Hypertension grades 2 and 3